CLINICAL TRIAL: NCT01670409
Title: A Phase II Study of Simultaneous Modulated Accelerated Radiation Therapy Concurrent With Chemotherapy in Patients With Esophageal Squamous Cell Carcinoma
Brief Title: Study of Simultaneous Modulated Accelerated Radiation Therapy Concurrent With Chemotherapy to Treat Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chuangzhen Chen (Other)
Responsible Party: Sponsor-Investigator, Chuangzhen Chen, M.D., Shantou University Medical College
Organization: Shantou University Medical College (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUMC-ECA-001; ChiCTR-ONC-12002356 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2012-08-12; First posted 2012-08-22 (Estimated); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Esophageal Neoplasms
Keywords: Esophageal squamous cell carcinoma; SMART; IMRT; Chemotherapy
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SMART combined with PF chemotherpay (Experimental): SMART-base IMRT with concurrent and adjuvant chemotherapy(cisplatin and 5-fluorouracil)
  Interventions: Radiation: SMART; Drug: PF

INTERVENTIONS:
Radiation: SMART — The PTV (planning target volume) of gross tumor will receive radiation dose of 66Gy, 2.2Gy per fraction and the PTV of subclinical disease will receive 54Gy, 1.8Gy per fraction,5 fraction per week.
Drug: PF — Concurrent and adjuvant chemotherapy: Cisplatin, 80mg/m2, intravenous on day 1, 5fluorouracil 0.5/m2, intravenous on d1 to d4. Two cycles during radiation treatment on d1 and d28. Two additional cycles after radiation treatment, 4 weeks per cycle.
  Other Names: cisplatin plus 5fluorouracil

SUMMARY:
The purpose of this study is to evaluate the acute and 2-year late toxicities, the 2-year local control and overall survival rates in patients with esophageal squamous cell carcinoma receiving simultaneous modulated accelerated radiation therapy concurrent with chemotherapy.

DETAILED DESCRIPTION:
Esophageal cancer is one of the most common malignant diseases in China, especially in Chaoshan region. Concurrent chemoradiotherapy is the standard non-surgical treatment method for this disease and the radiation schedule is about 50.4~60 Gray (Gy) in total, 1.8~2Gy per fraction generally. However, although with such comprehensive method, noncontrol of local disease or recurrence is still the main reason of failure.

Most patients with esophageal cancer suffer from malnutrition. A number of factors including hypoxic, inflammation, radioresistance and accelerated repopulation may contribute to local failures of disease after treatment; therefore a higher radiation biological equivalent dose (BED) will improve the local control probability. Although the intergroup 0123 (INT123) trial had shown that simply increasing total radiation dose could not gain better local control or overall survival rate, however, the ability of this trial to test the potential benefits of higher radiation dose could be compromized by the deficiencies within them, such as, observation bias,large radiated target volume and usage of conventional radiation technique. In other words, the probability that increasing radiation may help improving the control of disease should not be denied.

Modern radiation techniques, such as intensity modulation radiation therapy (IMRT), specially, are able to improve the coverage of target volumes and sparing of critical structures, while increase the total radiation dose. By using simultaneous modulated accelerated radiation therapy (SMART) technique, the doses to the relevant normal organs per fraction could be reduced significantly, while the doses to tumor could be increased to higher than 2Gy. Thus reach the double goal of protection of normal tissues, increasing total radiation Equivalent Uniform Dose (EUD). Dosimetric study has proven the feasibility and superiority of SMART-base IMRT in radiation treatment of esophageal cancer, compared with conventional technique.

Overall, SMART-base IMRT concurrent with chemotherapy may improve the local control and overall survival rate of patients with esophageal cancer; Meanwhile, the acute and late toxicities would be tolerable and slighter than that of conventional technique.

ELIGIBILITY:
Inclusion Criteria:

* pathological proven diagnosis of primary squamous cell carcinoma of the esophagus
* the primary disease located in cervical, upper or middle thoracic esophagus
* no distant metastases
* zubrod performance status: 0~2
* life expectancy > 6 months; -absence of another malignancy
* adequate liver, renal and bone marrow function
* women of childbearing potential and male participants must practice adequate contraception
* patient must provide study-specific informed consent prior to study entry

Exclusion Criteria:

* evidence of tracheoesophageal or Mediastinal-esophageal fistula
* prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years
* prior radiation therapy that would result in overlap of planned radiation therapy fields; - Severe, active comorbidity
* pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
* women who are nursing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Toxicities | The period during treatment and the 2 years after treatment
  The probabilities of grade ≥ 3 acute toxicities and 2-year late toxicities of esophagus and lungs as assessed by CTCAE 4.0

SECONDARY OUTCOMES:
Local control rate | 2 years after treatment
  The percentage of patients without locoregional tumor recurrence 2 years after treatment
overall survival rate | 2 years after treatment
  The percentage of patients that are alive 2 years after treatment
Complete blood count | before radiation treatment and after every 5 fraction of radiotherapy (7 time points in total)
  The complete blood count as assessed by a Coulter (LH 750 Haematology Analyzer)

CONTACTS AND LOCATIONS:
Overall Officials: Chuangzhen Chen, MD, Principal Investigator — Cancer Hospital, Shantou University Medical College
Locations (1):
- Cancer Hospital, Shantou University Medical College, Shantou, Guangdong, China

REFERENCES:
- [Derived] Liu W, Zeng C, Wang S, Zhan Y, Huang R, Luo T, Peng G, Wu Y, Qiu Z, Li D, Wu F, Chen C. A combined predicting model for benign esophageal stenosis after simultaneous integrated boost in esophageal squamous cell carcinoma patients (GASTO1072). Front Oncol. 2022 Dec 22;12:1026305. doi: 10.3389/fonc.2022.1026305. eCollection 2022. PMID 37078004
- [Derived] Zhang WZ, Chen JZ, Li DR, Chen ZJ, Guo H, Zhuang TT, Li DS, Zhou MZ, Chen CZ. Simultaneous modulated accelerated radiation therapy for esophageal cancer: a feasibility study. World J Gastroenterol. 2014 Oct 14;20(38):13973-80. doi: 10.3748/wjg.v20.i38.13973. PMID 25320535